CLINICAL TRIAL: NCT06780800
Title: Validity, Reliability, and Cross-Cultural Adaptation of the Turkish Version of Back Pain Knowledge and Beliefs Survey (BacKS)
Brief Title: Turkish Version of Back Pain Knowledge and Beliefs Survey
Acronym: BacKS-tr
Status: Active, not recruiting | Type: Observational
Sponsor: Ordu University (Other)
Collaborators: Macquarie University, Australia (Other)
Responsible Party: Principal Investigator, FUAT YUKSEL, Principal Investigator, Ordu University
Other Study IDs: E-14647249-000-1075264
Record Dates: First submitted 2025-01-06; First posted 2025-01-17 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Back Pain; Knowledge; Beliefs; Translation, Cultural Adaptation and Turkish Validation
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Test-retest group: One hundred of the participants who were administered the Tr-BacKS will fill out the same form again after 1 week.
  Interventions: Other: Backs-tr retest
- Test group: The questionnaire will be administered once to these 100 participants
  Interventions: Other: The Back Belief Questionnaire Tr (BBQ) and Backs-tr

INTERVENTIONS:
Other: The Back Belief Questionnaire Tr (BBQ) and Backs-tr — 200 people will be administered The Back Belief Questionnaire Tr (BBQ) and Backs-tr.
  Groups: Test group
Other: Backs-tr retest — 100 people will fill in the Backs-tr again after 1 week.
  Groups: Test-retest group

SUMMARY:
Low back pain (LBP) is a globally prevalent health issue, affecting the majority of individuals at some point in their lives. Misconceptions about LBP can prolong its chronicity, highlighting the importance of educating patients with accurate information. The Back Pain Knowledge and Beliefs Survey (BacKS), introduced in 2024, aims to measure individuals' knowledge about LBP based on updated scientific evidence. Given the high prevalence of LBP in Turkey and the lack of validated tools in Turkish, adapting BacKS to Turkish is essential. This study aims to conduct its cross-cultural adaptation, validation, and reliability analysis for clinical and community use.

DETAILED DESCRIPTION:
Low back pain (LBP) is one of the most prevalent health issues worldwide, with approximately three-quarters of individuals experiencing this condition at some point in their lives. Misconceptions, beliefs, and misinformation about LBP can prolong the duration of pain and contribute to its chronicity. Clinical guidelines emphasize the importance of educating patients with evidence-based information to remove potential barriers to recovery.

The Back Pain Knowledge and Beliefs Survey (BacKS) was introduced in October 2024 to assess individuals' knowledge and beliefs about LBP based on the most recent scientific evidence. Several tools in the literature aim to measure knowledge and beliefs related to LBP, including the Back Beliefs Questionnaire (BBQ) and the Back Pain Knowledge Questionnaire. However, these tools were developed in previous decades and may not reflect the current scientific literature. Additionally, the Turkish versions of some of these questionnaires have not yet undergone validation and reliability studies.

According to the 2016-2022 Turkish Health Survey conducted by the Turkish Statistical Institute (TÜİK), back-related problems rank first among all reported health issues, with a prevalence rate of 24.6%. Despite the high prevalence of LBP in Turkey, there is currently no systematically validated tool available in Turkish to measure the public's knowledge and beliefs regarding this condition.

The adaptation of BacKS into Turkish will help address this gap by providing a valid and reliable tool for both clinical and community-based research. Measuring and evaluating patient-reported outcomes accurately is crucial in managing LBP effectively. Therefore, the aim of this study is to conduct the cross-cultural adaptation, validation, and reliability analysis of the Turkish version of BacKS.

ELIGIBILITY:
Inclusion Criteria:

* Having low back pain or having a history of low back pain in the last 12 months
* To be able to read and write Turkish

Exclusion Criteria:

* Having cognitive impairment that prevents communication
* Pregnancy
* Malignite
* Infections
* Fractures,
* Inflammatory diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with current low back pain or a history of low back pain in the last 12 months.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Validation | 15.01.2025- 15.04.2025
  200 people will be compared with the scores obtained from the Backs-Tr questionnaire
The Back Belief Questionnaire (BBQ). | 15.01.2025- 15.04.2025
  200 people will be compared with the scores obtained from The Back Belief Questionnaire (BBQ).

SECONDARY OUTCOMES:
Reliability | 15.01.2025- 15.04.2025
  One hundred of the participants who were administered the Tr-BacKS will fill out the same form again after 1 week. The two measurement scores obtained from the participants will be compared using the Intraclass Correlation Coefficient (ICC).
Internal Consistency Reliability | 15.01.2025- 15.04.2025
  Internal consistency will be assessed separately for the biomedical (9 items) and self-care factor (11 items) in the original questionnaire. Internal consistency reliability will also be assessed for all items. Cronbach's Alpha will be used in the evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Ordu University, Ordu, altinordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No